CLINICAL TRIAL: NCT05593887
Title: Late-presenting Hip Dislocation in Non-ambulatory Children With Cerebral Palsy: A Comparison of Three Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Ayoub (Other)
Responsible Party: Sponsor-Investigator, Muhammad Ayoub, Principle Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cp dislocated hip
Record Dates: First submitted 2022-10-17; First posted 2022-10-26 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral palsy; McHale; dislocated hip; GMFCS IV; GMFCS V; Hip reconstruction surgery; HRS; Proximal femoral resection; valgus osteotomy
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hip Reconstruction surgery. (Active Comparator): This group will undergo Hip reconstruction surgery Anterior approach overlying the iliac crest: open reduction and pelvic osteotomy. Lateral approach: derotation-varization osteotomy and shortening of femur and internal fixation.
  Interventions: Procedure: Hip reconstruction surgery.
- Proximal femoral resection (Active Comparator): This group will undergo PFR as described by resection of the proximal part of the femur below the level of the lesser trochanter by 2 to 3 cm and constructed a capsular flap across the acetabulum. The quadriceps muscle will be sutured around the resected end of the femur.
  Interventions: Procedure: Proximal femoral resection
- Proximal femur valgus osteotomy (Active Comparator): This group will undergo McHale Procedure.The patient is positioned in the lateral decubitus Position A straight incision is cantered over the greater trochanter and extends proximally. Head and neck are resected. A closing wedge, shortening, valgus-producing osteotomy of 40 to 50 degrees is marked just below the lesser trochanter and fixed by a plate.
  Interventions: Procedure: Proximal femoral valgus ostetomy

INTERVENTIONS:
Procedure: Hip reconstruction surgery. — This group will undergo Hip reconstruction surgery Anterior approach overlying the iliac crest: open reduction, pelvic osteotomy and pelvic osteotomy. Lateral approach: derotation-varization osteotomy and shortening of femur, internal fixation
  Other Names: Varus derotation shortening ostetomy.
  Arms: Hip Reconstruction surgery.
Procedure: Proximal femoral resection — Resection of the proximal part of the femur below the level of the lesser trochanter by 2 to 3 cm and constructed a capsular flap across the acetabulum. The quadriceps muscle will be sutured around the resected end of the femur
  Other Names: Castle shnider procedure
  Arms: Proximal femoral resection
Procedure: Proximal femoral valgus ostetomy — The patient is positioned in the lateral decubitus Position A straight incision is cantered over the greater trochanter and extends proximally. Head and neck are resected. A closing wedge, shortening, valgus-producing osteotomy of 40 to 50 degrees is marked just below the lesser trochanter and fixed by a plate
  Other Names: McHale procedure
  Arms: Proximal femur valgus osteotomy

SUMMARY:
Cerebral palsy (CP) is characterized by a fixed lesion that affects the neurological system during development. Pathologic hip conditions, such as subluxation or dislocation, are of great concern in non-ambulatory CP patients. Complete hip dislocations are commonly encountered in non-ambulatory CP patients and this can be quite problematic if pain is experienced or when sitting, balance, posture, or hygiene become affected.

The management of this patient population includes both reconstructive surgery, which aimed to center the dislocated femoral head into the acetabulum, and salvage surgeries, which are performed to reduce associated pain and/or functional deficits (e.g., sitting problems).

There are many options for salvage management of dislocated hips in CP patients, including proximal femoral resection (PFR) either with or without cartilage capping, proximal femoral valgus osteotomy, hip arthrodesis, and prosthetic hip arthroplasty.

To date, there is no conclusive evidence to determine which option is superior compared to the others in terms of efficacy and postoperative complications in CP patients due to the lack of a comparison group and the small number of included patients. Furthermore, the decision to take reconstructive vs. salvage procedures is still a matter of debate in the literature.

Therefore, this study is being conducted to compare outcomes between PFR, reconstructive hip surgery, and proximal femur valgus osteotomy in terms of clinical improvement (Including pain) and complications

DETAILED DESCRIPTION:
Hip displacement is common in non-ambulatory patients with cerebral palsy (CP) of Gross Motor Function Classification System (GMFCS) levels IV and V. CP is a permanent disorder affecting movement and posture that causes activity limitations due to nonprogressive injury to the fetal or immature infant brain. Owing to the primary abnormalities of CP, such as spasticity and muscle imbalance, hip displacement progresses and is usually detected around the age of five to seven years old. If left untreated, progressive hip displacement eventually causes pain, pelvic obliquity, difficulty with sitting, and hinders hygiene.

Neglected dislocation leads to femoral head deformity and it is assessed with the use of the revised version of the MCPHCS (Melbourne Cerebral Palsy Hip Classification system). The MCPHCS is a radiographic classification system that includes joint congruency and alignment as well as acetabular and femoral head deformity.

Previous studies have shown that reduction of displacement through hip reconstructive surgery (HRS), which includes femoral varus and de-rotational osteotomy (FVDO), with or without pelvic osteotomies, relieves both pain frequency and intensity

. It has been found however that hip joint congruity after HRS improves even if the initial presentation of a CP hip seems irreversible.

There are many options for salvage management of dislocated hips in CP patients, including proximal femoral resection (FHR) either with or without cartilage capping, which is known as femoral head cap plastic surgery (FCP), and proximal femoral valgus osteotomy.

Noteworthy, pain and muscular spasm are frequent postoperative complaints during the early postoperative period, particularly before the benefits of FCP and FHR can be witnessed. Thus, a number of management strategies can be used to control these symptoms, including the use of analgesics, anxiolytics, or skin traction.

Horsch et al in their study found that the postoperative outcomes of FHR and FCP are similar in terms of telescoping, heterotopic ossification, and complication.

Traditionally, resection arthroplasty has been considered as an option for palliative treatment of a CP hip with femoral head destruction. However, there are no clear-cut indications for resection arthroplasty for a deformed femoral head.

The procedure described by McHale in 1990 entails femoral head and neck resection, valgus-producing subtrochanteric osteotomy to reposition the leg relative to the trunk, and advancement of the lesser trochanter into the acetabulum by attaching ligamentum teres to the intact iliopsoas. To date, there is no conclusive evidence to determine which option is superior compared to the others in terms of efficacy and postoperative complications in CP patients due to the lack of a comparison group, the small number of included patients, and the short follow-up periods. Therefore, A prospective study will be conducted to compare outcomes between Proximal femoral resection (Castle Schneider), Valgus osteotomy (McHale procedure), and Reconstructive hip procedure (VDO + Pelvic osteotomy) as regards post-operative clinical and radiological changes and postoperative complications that include pain, proximal migration, stiffness, and Heterotrophic ossifications.

ELIGIBILITY:
Inclusion Criteria:

* Lesion: neglected deformed dislocated hip (Deformed head Group B, C, and D according to Rutz classification modified from MCPHCS )
* Non-ambulatory: as defined by GMFCS level IV and V

Exclusion Criteria:

* Ambulatory patients
* patients underwent any previous hip bony procedures.
* Non-deformed Femoral head Group A according to Rutz classification
* Neuromuscular hip dislocation other than cp.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-10-26 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Radiological changes | Immediately postoperative, 3 weeks postoperative, 3 months postoperative, and 6 months postoperative
  Plain radiograph x-ray is used to assess the Migration percentage
Radiological changes | Immediately postoperative, 3 weeks postoperative, 3 months postoperative, and 6 months postoperative
  Plain radiograph x-ray is used to assess Pelvic obliquity
Radiological changes | Immediately postoperative, 3 weeks postoperative, 3 months postoperative, and 6 months postoperative
  Plain radiograph x-ray is used to asses Acetabular index.
Radiological changes | Immediately postoperative, 3 weeks postoperative, 3 months postoperative, and 6 months postoperative
  Plain radiograph x-ray is used to assess Femoral head sphericity
Radiological changes | Immediately postoperative, 3 weeks postoperative, 3 months postoperative, and 6 months postoperative
  Plain radiograph x-ray is used to assess Femoral head deformity.
Radiological changes | Immediately postoperative, 3 weeks postoperative, 3 months postoperative, and 6 months postoperative
  Plain radiograph x-ray is used to assess Proximal Femoral Migration.
Radiological changes | Immediately postoperative, 3 weeks postoperative, 3 months postoperative, and 6 months postoperative
  Plain radiograph x-ray is used to assess Heterotrophic ossification
Clinical changes | 6 weeks post operative, 3 months postoperative, and 6 months postoperative
  Cp quality of life Questionnaire ( preoperative and postoperative). No minimum or maximum score. Increase score means clinical improvement.
Clinical changes | 6 weeks post operative, 3 months postoperative, and 6 months postoperative
  Non-communicating children's pain checklist - revised ( preoperative and postoperative).score equals or more than 7 indicates that the child is in pain. Increase score means more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mootaz Thakeb, MD, Study Chair — Ain Shams University
Locations (1):
- Faculty of medicine, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terjesen T. Development of the hip joints in unoperated children with cerebral palsy: a radiographic study of 76 patients. Acta Orthop. 2006 Feb;77(1):125-31. doi: 10.1080/17453670610045803. PMID 16534712
- [Background] Lins LAB, Watkins CJ, Shore BJ. Natural History of Spastic Hip Disease. J Pediatr Orthop. 2019 Jul;39(Issue 6, Supplement 1 Suppl 1):S33-S37. doi: 10.1097/BPO.0000000000001347. PMID 31169645
- [Background] DiFazio R, Shore B, Vessey JA, Miller PE, Snyder BD. Effect of Hip Reconstructive Surgery on Health-Related Quality of Life of Non-Ambulatory Children with Cerebral Palsy. J Bone Joint Surg Am. 2016 Jul 20;98(14):1190-8. doi: 10.2106/JBJS.15.01063. PMID 27440567
- [Background] Robin J, Graham HK, Baker R, Selber P, Simpson P, Symons S, Thomason P. A classification system for hip disease in cerebral palsy. Dev Med Child Neurol. 2009 Mar;51(3):183-92. doi: 10.1111/j.1469-8749.2008.03129.x. Epub 2008 Dec 3. PMID 19055594
- [Background] Braatz F, Eidemuller A, Klotz MC, Beckmann NA, Wolf SI, Dreher T. Hip reconstruction surgery is successful in restoring joint congruity in patients with cerebral palsy: long-term outcome. Int Orthop. 2014 Nov;38(11):2237-43. doi: 10.1007/s00264-014-2379-x. Epub 2014 Jun 27. PMID 24968787
- [Background] Min JJ, Kwon SS, Sung KH, Lee KM, Chung CY, Park MS. Remodelling of femoral head deformity after hip reconstructive surgery in patients with cerebral palsy. Bone Joint J. 2021 Jan;103-B(1):198-203. doi: 10.1302/0301-620X.103B1.BJJ-2020-1339.R1. PMID 33380203
- [Background] Shaw KA, Hire JM, Cearley DM. Salvage Treatment Options for Painful Hip Dislocations in Nonambulatory Cerebral Palsy Patients. J Am Acad Orthop Surg. 2020 May 1;28(9):363-375. doi: 10.5435/JAAOS-D-19-00349. PMID 31663909
- [Background] Dartnell J, Gough M, Paterson JM, Norman-Taylor F. Proximal femoral resection without post-operative traction for the painful dislocated hip in young patients with cerebral palsy: a review of 79 cases. Bone Joint J. 2014 May;96-B(5):701-6. doi: 10.1302/0301-620X.96B5.32963. PMID 24788508
- [Background] Horsch A, Hahne F, Ghandour M, Platzer H, Alimusaj M, Putz C. Radiological Outcomes of Femoral Head Resection in Patients with Cerebral Palsy: A Retrospective Comparative Study of Two Surgical Procedures. Children (Basel). 2021 Dec 1;8(12):1105. doi: 10.3390/children8121105. PMID 34943303
- [Background] McHale KA, Bagg M, Nason SS. Treatment of the chronically dislocated hip in adolescents with cerebral palsy with femoral head resection and subtrochanteric valgus osteotomy. J Pediatr Orthop. 1990 Jul-Aug;10(4):504-9. PMID 2358491
- [Background] Rutz E, Vavken P, Camathias C, Haase C, Junemann S, Brunner R. Long-term results and outcome predictors in one-stage hip reconstruction in children with cerebral palsy. J Bone Joint Surg Am. 2015 Mar 18;97(6):500-6. doi: 10.2106/JBJS.N.00676. PMID 25788307
- [Background] Waters E, Maher E, Salmon L, Reddihough D, Boyd R. Development of a condition-specific measure of quality of life for children with cerebral palsy: empirical thematic data reported by parents and children. Child Care Health Dev. 2005 Mar;31(2):127-35. doi: 10.1111/j.1365-2214.2004.00476.x. PMID 15715691
- [Background] Breau LM, McGrath PJ, Camfield CS, Finley GA. Psychometric properties of the non-communicating children's pain checklist-revised. Pain. 2002 Sep;99(1-2):349-57. doi: 10.1016/s0304-3959(02)00179-3. PMID 12237214
- [Background] Shrader MW, Andrisevic EM, Belthur MV, White GR, Boan C, Wood W. Inter- and Intraobserver Reliability of Pelvic Obliquity Measurement Methods in Patients With Cerebral Palsy. Spine Deform. 2018 May-Jun;6(3):257-262. doi: 10.1016/j.jspd.2017.10.001. PMID 29735134